CLINICAL TRIAL: NCT04692194
Title: Study "HEMORROIDAL SURGERY AND Chronic Inflammatory Bowel Disease"
Acronym: CHRMICI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CHRMICI
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hemorrhoids; Chronic Inflammatory Bowel Disease
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemorrhoidal surgery is considered potentially harmful in patients with chronic inflammatory bowel disease (IBD). Patients with Crohn's disease may have ano-perineal involvement during the course of the disease or even before diagnosis. In addition, patients with IBD (Crohn's or RectoColitis Haemorrhagic, UC) may have rectal involvement. In both cases, hemorrhoidal surgery can be harmful to the anorectal level. However, recent data from the literature has proven to be reassuring. Indeed, the latest studies published on this subject have shown that hemorrhoidal surgery can be performed in a large majority of patients with IBD, especially when the disease is quiescent.

The main objective is to assess the morbidity of hemorrhoidal surgery in IBD patients who have been operated on at our center. Postoperative complications will be the main elements sought in the study.

The secondary objective is to search for predictive factors of complications from hemorrhoidal surgery in patients with IBD. This requires an exhaustive collection of clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient with IBD (Crohn's or UC) with a diagnosis prior to hemorrhoidal surgery
* Patient operated on for hemorrhoidal surgery performed between November 1, 2013 and July 7, 2020 in our center
* French-speaking patient

Exclusion Criteria:

* Patient with severe inflammatory disease
* Patient with ano-perineal involvement of Crohn's disease
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Patient objecting to the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with IBD (Crohn's or UC) with a diagnosis prior to hemorrhoidal surgery, operated on for hemorrhoidal surgery performed between November 1, 2013 and July 7, 2020 in our center
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Morbidity from hemorrhoidal surgery | Year 1
  This outcome corresponds to the prevalence of postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Amine ALAM, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Groupe Hospitalier Paris Saint-Joseph, France

REFERENCES:
- [Result] Cracco N, Zinicola R. Is haemorrhoidectomy in inflammatory bowel disease harmful? An old dogma re-examined. Colorectal Dis. 2014 Jul;16(7):516-9. doi: 10.1111/codi.12555. PMID 24422778
- [Result] Jeffery PJ, Parks AG, Ritchie JK. Treatment of haemorrhoids in patients with inflammatory bowel disease. Lancet. 1977 May 21;1(8021):1084-5. doi: 10.1016/s0140-6736(77)92337-6. PMID 68184
- [Result] McKenna NP, Lightner AL, Habermann EB, Mathis KL. Hemorrhoidectomy and Excision of Skin Tags in IBD: Harbinger of Doom or Simply a Disease Running Its Course? Dis Colon Rectum. 2019 Dec;62(12):1505-1511. doi: 10.1097/DCR.0000000000001524. PMID 31580261
- [Result] Lightner AL, Kearney D, Giugliano D, Hull T, Holubar SD, Koh S, Zaghiyan K, Fleshner PR. Excisional Hemorrhoidectomy: Safe in Patients With Crohn's Disease? Inflamm Bowel Dis. 2020 Aug 20;26(9):1390-1393. doi: 10.1093/ibd/izz255. PMID 31633186